CLINICAL TRIAL: NCT00884975
Title: Exacerbations and Health Related Quality of Life in Chronic Obstructive Pulmonary Disease: CRECOPD Study
Brief Title: Exacerbations and Health Related Quality of Life in Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Demosthenes Makris, University of Thessaly
Other Study IDs: DM19021970DM
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; exacerbations; quality of life; emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic obstructive pulmonary disease (COPD) exacerbation is a major cause of physician visits and hospital admissions associated with acute respiratory failure, causing increased morbidity and premature mortality and thus it can significantly affect Health Related Quality of Life (HRQoL).

Previous studies suggested that patients who have experienced frequent exacerbation present worse HRQoL compared to patients with infrequent exacerbations. However, there are still questions regarding the relationship between HRQoL and exacerbations.

In the present study the investigators will study a cohort of COPD patients over 6 years, they will document exacerbations, they will assess lung emphysema by computed tomography of the chest and they will evaluate health related quality of life in COPD patients.

The investigators hypothesize that the extend of emphysema in COPD patients is positively correlated with worsen Health related quality of life (HRQoL).

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is characterized by progressive loss of lung function and recurrent exacerbations. COPD exacerbation is a major cause of physician visits and hospital admissions associated with acute respiratory failure, causing increased morbidity and premature mortality and thus it can significantly affect HRQoL.

Previous studies suggested that patients who have experienced frequent exacerbation present worse HRQoL compared to patients with infrequent exacerbations. However, there are still questions regarding the relationship between HRQoL and exacerbations. Only few studies which are not an integral part of a clinical trial investigated the relationship between exacerbations and long-term impairment of HRQoL. Furthermore, a recent study failed to show that exacerbations remain a significant determinant of HRQoL when several other prognostic factors were taken into account. In addition, there is luck of data regarding differences in HRQoL between patients with different phenotypes (i.e., emphysema or chronic bronchitis predominance).

In this respect we prospectively study the long term effect of exacerbations on the quality of life of patients with COPD and we aim to investigate further the relationship between exacerbations and HRQoL.

The investigators hypothesize that the extend of emphysema is positively correlated with worsen Health related quality of life (HRQoL).

Consecutive sampling will be used to recruit patients with a diagnosis of COPD according to the GOLD definition.Exacerbations will be identified as worsening of patient's respiratory signs as recorded on diary cards. HQoL will be assessed using the Saint George Respiratory Questionaire (SGRQ). Patients will undergo high resolution computed tomography of the chest(HRCT). Multiple linear regression analysis will be used to identify factors which explain SGRQ deterioration over the study period for the entire population and for smokers and ex-smokers separately.

ELIGIBILITY:
Inclusion Criteria:

* chronic Obstructive Lung Disease diagnosis
* ability to perform spirometry

Exclusion Criteria:

* previously diagnosed or clinically evident bronchiectasis
* history of Asthma or other respiratory disease
* continuous use of systemic steroids more than 30 days in the previous year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Chronic Obstructive Lung Disease according to the GOLD definition (Pauwels RA, Buist AS, Calverley PM, et al; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001;163(5):1256-76.), who attend outpatient clinics at Chania General Hospital on the island of Crete, Greece
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2002-05; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Demos Makris, MD, Principal Investigator — University of Crete/University of Thessaly